CLINICAL TRIAL: NCT00654108
Title: A Randomized, Double-Blind, Placebo-Controlled Dose Escalation, Inpatient Phase I Study to Determine the Safety and Immunogenicity of a Single Oral Dose of a Combined Live, Attenuated, Enterotoxigenic Escherichia Coli (ETEC)-Cholera Vaccine (Peru-15 pCTB) in Healthy Adult Subjects
Brief Title: Safety and Immunogenicity of Peru-15-pCTB in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 07-0052
Record Dates: First submitted 2008-04-03; First posted 2008-04-07 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2010-02-09

CONDITIONS: Gastroenteritis Escherichia Coli
Keywords: cholera; diarrhea; Escherichia coli; vaccine
MeSH Terms: conditions — Cholera; Diarrhea; Escherichia coli Infections | interventions — Ciprofloxacin; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1: vaccine dosage level 1 or placebo (Experimental): Vaccine dose level 1: 1 X 10^7 colony forming unit (CFU) or placebo, treated with Cipro on days 7-11.
  Interventions: Drug: Ciprofloxacin; Biological: Peru-15-pCTB; Other: Sodium bicarbonate/Ascorbic Acid/Aspartame Buffer
- Cohort 2: vaccine dosage level 2 or placebo (Experimental): Vaccine dose level 2: 1 X 10^8 CFU or placebo, treated with Cipro on days 7-11.
  Interventions: Drug: Ciprofloxacin; Biological: Peru-15-pCTB; Other: Sodium bicarbonate/Ascorbic Acid/Aspartame Buffer
- Cohort 3: vaccine dosage level 3 or placebo (Experimental): Vaccine dose level 3: 1 X 10^9 CFU or placebo, treated with Cipro on days 7-11.
  Interventions: Drug: Ciprofloxacin; Biological: Peru-15-pCTB; Other: Sodium bicarbonate/Ascorbic Acid/Aspartame Buffer
- Cohort 4: vaccine dosage level 4 or placebo (Experimental): Vaccine dose level 4: 1 X 10^10 CFU or placebo, treated with Cipro on days 7-11.
  Interventions: Drug: Ciprofloxacin; Biological: Peru-15-pCTB; Other: Sodium bicarbonate/Ascorbic Acid/Aspartame Buffer

INTERVENTIONS:
Drug: Ciprofloxacin — 500 milligrams(mg) will be administered orally twice daily for 5 days.
Biological: Peru-15-pCTB — Live attenuated oral combined ETEC-cholera (Peru-15 pCTB) vaccine co-administered with bicarbonate buffer solution; vaccine dose levels 1 X 10^7; 1 X 10^8; 1 X 10^9; and 1 X 10^10.
Other: Sodium bicarbonate/Ascorbic Acid/Aspartame Buffer — Buffer solution: 2.5 grams (g) Sodium Bicarbonate powder, 1.65 g Ascorbic Acid and 25 mg Aspartame, in 100 milliliters (mL) water for injection.

SUMMARY:
Enterotoxigenic Escherichia (E.) coli (ETEC) bacteria are the main cause of traveler's diarrhea and are significant pathogens affecting children and elderly individuals of developing countries. The purpose of the study is to determine the safety of the ETEC-Cholera vaccine and the body's ability to protect itself against ETEC and cholera infection after receiving the vaccine. The study will enroll a total of 64 healthy volunteers, 18 to 45 years old at the Cincinnati Children's Hospital. The study will provide increasing doses of the vaccine or placebo (inactive substance) to 4 groups consisting of 16 participants each. Participants will remain in the inpatient unit for observation for about 11 days. All subjects will be treated with Cipro, an antibiotic, for 5 days. Study procedures include: blood samples, vital signs, physical examinations, and stool samples. Volunteers will be involved in the study for about 8 months including telephone contacts.

DETAILED DESCRIPTION:
Enterotoxigenic Escherichia coli (ETEC) are the principal single cause of traveler's diarrhea and are a significant pathogen affecting children and elderly individuals of developing countries. ETEC infections result in approximately 600 million total cases of diarrhea worldwide annually, with an estimated 280 million cases and over 400,000 deaths in children less than 5 years of age. The proposed study is a randomized, double-blind, placebo controlled, dose-escalation, inpatient Phase I study to determine the safety and immunogenicity of a single oral dose of a combined live, attenuated, enterotoxigenic Escherichia coli (ETEC)-cholera vaccine (Peru-15 pCTB). A total of 64 healthy subjects, 18 to 45 years old will be enrolled in this study. Subject participation duration is up to 8 months. Sequential cohorts of 16 eligible subjects will be randomized in a 3:1 ratio to receive the assigned dose of ETEC-cholera vaccine or placebo (bicarbonate buffer only), respectively. The first dose level cohort (1x10^7 colony forming units) will be divided into 2 groups. Initially, 4 subjects will be enrolled, treated, and observed to ensure the tolerability of this dose level through Day 28. In the absence of any stopping rules, enrollment and dosing will proceed with the remaining 12 subjects of this cohort. Thereafter, dose escalation and subject enrollment will proceed in a step-wise fashion. A Safety Monitoring Committee will be convened for this study, and will review available safety data through the Day 28 post-vaccination visits for each cohort prior to making a recommendation to the Sponsor on advancement to the next dose level. The study will be conducted at Cincinnati Children's Hospital. The primary objective of this study will be to assess the safety of a combined ETEC-cholera vaccine [Peru-15-pCTB (Cholera toxin B-subunit)] when administered as a single oral dose over a range of doses in healthy adult subjects compared to placebo at day 28 post-vaccination. The secondary objectives will be: to assess long-term safety follow-up from immunization through Month 6 post vaccination; to evaluate the immunogenicity of a single oral dose of ETEC-cholera vaccine over a range of doses in healthy adult subjects; and to evaluate the shedding profile of the ETEC-cholera vaccine organisms in stool for a period of 7 days.

ELIGIBILITY:
Inclusion Criteria:

-Male or female age 18-45, inclusive. -Healthy as judged by the Principal Investigator (PI) and determined by medical history, physical examination, vital signs, screening laboratories, and medication history. -Capable of understanding, consenting and complying with the entire study protocol including the inpatient period. -Female subjects must be of non-childbearing potential, or if of childbearing potential (as determined by the investigator) must be practicing abstinence or using an effective licensed method of birth control (e.g., oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream, or foam; intrauterine contraceptive device, or Depo-Provera; skin patch; vaginal ring or cervical cap) for 30 days prior to vaccination and must agree to continue such precautions during the study and for 30 days after the Day 28 study visit. -Male subjects must agree not to father a child during the study and for 90 days after the Day 0 study visit. -Provide voluntary written informed consent and attained at least 70% on an examination about the study on the first attempt. -Have normal screening laboratories for serum glutamic pyruvic transaminase (SGPT) alanine aminotransferase (ALT), creatinine, sodium, potassium, total white blood count (WBC), hemoglobin, neutrophils, lymphocytes, platelets, urine protein, urine glucose and urine red blood cells (RBC).

Exclusion Criteria:

-Women who are pregnant or lactating or have a positive serum pregnancy test at screening or upon admission to inpatient facility. -Subjects who are immunocompromised or immunodeficient, or have had a prior malignancy (exception: a history of basal cell or squamous cell carcinoma in remission without treatment for more than 5 years prior to study entry). -History of clinically significant chronic illness or other condition requiring chronic medication therapy. -History of malabsorption or maldigestion disorder (e.g., celiac sprue), major gastrointestinal (GI) surgery, or any other chronic GI disorders that would interfere with the study or the investigational product. -Any current or past use of immunosuppressive medications including inhaled steroids (e.g., for asthma) within 6 months of screening. -Recent (e.g., within 5 years) history of travel to a cholera or Enterotoxigenic Escherichia coli (ETEC) endemic area, raised in a cholera or ETEC endemic area or a history of raising a child from an endemic area for cholera or ETEC. Individuals who may work with Vibrio (V) cholerae or ETEC in the laboratory are also excluded. -Vaccination against or infection with cholera or E. coli, or participation in a clinical trial using cholera or ETEC vaccine or organisms at any time. -History of drug or alcohol abuse any time in the last 6 months. -Presence of HIV antibody, hepatitis C antibody, or positive hepatitis B surface antigen. -Clinically abnormal screening electrocardiogram (ECG) defined as pathologic Q waves and significant ST-T wave changes; criteria for left ventricular hypertrophy; and any non-sinus rhythm excluding isolated premature atrial contractions. -Presence of bacterial or parasitic pathogens in stool culture in a screening stool examination. -IgA (immunoglobulin) deficiency. -A change in subject's normal stool pattern within 3 months of screening visit. A normal stool pattern is defined as 3 to 21 stools per week. -Any known allergy or sensitivity to Ciprofloxacin. -Have any known allergy to components of the vaccine [M9 minimal salts, glycerin, dextrose anhydrous, sodium chloride, peptone (vegetable) acid hydrolysate, magnesium sulfate heptahydrate, and aspartame] or placebo/bicarbonate buffer (water, sodium bicarbonate, ascorbic acid, and aspartame). -Any medical illness requiring a new prescription medication or hospitalization during the screening period or having a temperature greater than or equal to 38.0 degrees Celsius during the 2 weeks prior to investigational product administration (Day 0). -Administration of any vaccine, licensed or investigational, or any investigational product within 30 days of investigational product administration (Day 0) or any plan for participation in another investigational trial during this study. -Use of antibiotics within 7 days of investigational product administration (Day 0). -Use of laxatives for hard or infrequent stools one or more times in a month in any of the 3 months prior to enrollment. -Use of any H2 receptor antagonists (e.g., Tagamet®, Zantac®, and Pepcid®), proton pump inhibitors (e.g., Prilosec® over the counter (OTC), Protonix®, and Prevacid®), or prescription acid suppression medication or OTC antacids within 72 hours of investigational product administration. -Use of prescription and OTC medications that contain acetaminophen, aspirin, ibuprofen, and other nonsteroidal anti-inflammatory drugs within 48 hours prior to investigational product administration. -Employment as a commercial food handler, day care worker, or health care worker involved in direct patient contact. Subjects with children less than 2 years old at home or with household contacts that are immunocompromised, pregnant or breast-feeding. -Any other condition or responsibili ty, such as a medical, psychiatric, or social condition or occupational responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to the subject's participation in the protocol or assessment of the investigational product. -Subjects who are unwilling or unable to cease smoking for the duration of the inpatient stay. -Subjects who are unable to pass a test that describes cholera and ETEC diarrhea and explains the requirements of the clinical trial. Subjects must score a minimum of 70 percent upon the first attempt. -Subjects will be excluded if their screening laboratory test results fall outside of the laboratory normal; however, transaminase levels [alanine aminotransferase (ALT)] and creatinine levels (Cr) below the lower limit of "normal" will not be an exclusion criterion. -Subjects with Phenylketonuria (PKU) will be excluded because the investigational product (vaccine) bicarbonate buffer contains aspartame.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2008-06-02 (Actual); Primary Completion 2010-05-30 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) will be graded according to standardized criteria. | Through the Day 28 post-vaccination visit.
Safety: physical examinations, interim medical history, solicited symptoms/subject memory aid, and laboratory evaluations. | Through the Day 28 post-vaccination visit.

SECONDARY OUTCOMES:
Immunogenicity will be assessed by changes in vibriocidal antibody titer, anti-Cholera toxin B-subunit antibody titer, and anti-Labile toxin antibody titer. | Days -1, 7, 10, 14, and 28.
Stool shedding of the vaccine organisms will be assessed by qualitative and quantitative cultures. | Qualitative: Days 1-10, 14, 21, 28: Quantitative: Days 1-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Chen WH, Garza J, Choquette M, Hawkins J, Hoeper A, Bernstein DI, Cohen MB. Safety and immunogenicity of escalating dosages of a single oral administration of peru-15 pCTB, a candidate live, attenuated vaccine against enterotoxigenic Escherichia coli and Vibrio cholerae. Clin Vaccine Immunol. 2015 Jan;22(1):129-35. doi: 10.1128/CVI.00560-14. Epub 2014 Nov 19. PMID 25410205